CLINICAL TRIAL: NCT04723134
Title: Development of a Novel Folic Acid Wound Dressing to Enhance Nitric Oxide Bioactivity Required for Diabetic Foot Ulcer Wound Healing
Brief Title: Evaluation of a Folic Acid Wound Treatment (FAWT) for Chronic, Early-Stage Diabetic Foot Ulcer (DFU) Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Boykin, MD (U.S. Federal Agency)
Collaborators: George Mason University (Other); Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Joseph Boykin, MD, Medical Director, Wound Healing Program, Hunter Holmes Mcguire Veteran Affairs Medical Center
Organization: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFU/FAWT-001(8)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Wound Healing; Folic Acid; DNA Methylation
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Folic Acid Wound Treatment (Active Comparator): Intervention - participants receiving 2.5% folinic acid wound treatment for daily treatment of chronic early stage diabetic foot ulcer wound. This will be applied daily to the study wound selected for monitoring.
  Interventions: Combination Product: Folinic acid calcium salt
- Placebo (Placebo Comparator): Intervention - participants receiving Placebo (PluroGel Burn and Wound Dressing) for daily treatment of chronic early stage diabetic foot ulcer wound. This will be applied daily to the study wound selected for monitoring.
  Interventions: Combination Product: Folinic acid calcium salt

INTERVENTIONS:
Combination Product: Folinic acid calcium salt — Folinic acid (2.5%) by combination with Placebo
  Other Names: Placebo; PluroGel Burn and Wound Dressing

SUMMARY:
This is a twelve-week single-center, randomized, double-blind, clinical study to evaluate the safety and efficacy of a folic acid wound treatment (FAWT) versus Placebo in the promotion of healing of chronic, early stage diabetic foot ulcer (ES-DFU) wounds. Male and female Veterans with type-2 diabetes mellitus and chronic ES-DFUs acceptable to the study inclusion/exclusion criteria will be considered for enrollment.

DETAILED DESCRIPTION:
This clinical study is a twelve-week single-center, randomized, double-blind evaluation of the safety and efficacy of a folic acid wound treatment (FAWT) versus Placebo in the promotion of healing of chronic (greater than 4-weeks), early stage diabetic foot ulcer (ES-DFU) wounds (PEDIS-Grade 1 or 2 Depth - wound above fascia without exposed muscle, tendon or bone). Study wound areas will be between 1.0 and 12.0 cm-square.

The chronic, non-healing DFU is a serious and common complication of diabetes. Chronic DFU complications are among the most frequent diabetes-related diagnoses for hospitalization and the leading cause of diabetes-associated lower limb amputations. Increased levels of the tumor suppressor protein p53 in wound keratinocytes from non-healing DFUs suggests increased cell death due to significant (p<0.05) transcription factor activation. Treatment with high dose folic acid (5mg/day) correlates to improved healing in ES-DFU wounds, perhaps by improving folate/methionine metabolism which provides support for DNA repair, the generation of reductive equivalents and regulates DNA methylation, an important epigenetic regulator of p53 transcription activity. Folinic acid calcium salt (calcium folinate) is the bioactive metabolite of folic acid that does not require reduction by dihydrofolate reductase (DHFR). In this study, FAWT (2.5-percent by weight) is provided by compounding 1.25-gms of folinic acid calcium salt with 50-gms of the Placebo (Plurogel Burn and Wound Dressing™, Medline Industries, Inc.). Experimental studies of topical folinic acid demonstrate significant improvements in wound healing parameters with decreased cellular markers of inflammation and increased active signaling of tissue repair. Topical administration of FAWT removes the potential for the adverse impact of high blood folate levels observed with oral high dose folic acid, that could include an increase in the occurrence of sub-classes of colon or prostate cancer.

The study hypothesis is that during a twelve-week evaluation period FAWT may provide significant (p<0.05) improvements, as compared to Placebo, in the rate of healing and complete closure (re-epithelialization) of chronic ES-DFU wounds.

The study will have two phases: Screening and Treatment.

The Screening Phase (first 4 weeks) is designed to determine if male and female Veterans selected as study participants are eligible to proceed to the Treatment Phase of the study. This phase consists of screening assessments that will include evaluation of the rate of study wound closure while the participants receive standard of care (SOC) therapy, including off-loading. SOC treatment will include wound cleansing and sharp debridement, fluorescent surveillance of wounds for microbial colonization and the management of infections. Participants observed with greater than 50-percent wound area reduction at the end of 4-weeks will be excluded from entering the Treatment Phase. Those observed with less than 50-percent wound area reduction and who continue to meet the inclusion/exclusion criteria will be allowed to enter the Treatment Phase of the study.

The Treatment Phase (12 weeks) will continue with assessments of the eligibility of the remaining study participants. Thirty study participants (n=30) selected after the four-week Screening Phase will be randomly assigned to either the FAWT or Placebo group of fifteen subjects each (n=15). Study participants and the treating staff members will be blinded to the treatment (FAWT or Placebo) being provided to each participant. During the Treatment Phase subjects will be evaluated every two weeks. These evaluations will include the collection of selected blood chemistries, assessment of ulcer wound healing, wound measurements and microbial surveillance using digital imaging. Paired marginal wound tissue biopsies (3-mm) will be obtained during two points of the Treatment Phase: 1) at the beginning of the Treatment Phase and 2) following the complete closure of the wound or after twelve weeks of Treatment. Study evaluations of the wound will continue until the wound is closed or at twelve weeks, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be male or female Veterans with T2DM managed with insulin and/or non-insulin therapy who have a chronic, non-healing DFU (wound age: at least 4-weeks) and who have signed an Institutional Review Board approved informed consent document.
* Study subject candidates (SC) - may present with multiple DFUs; however, only one DFU per SC will be selected for study. A DFU-SC must be observed with: 1) at least a four-week history of a non-healing, superficial DFU-wound; PEDIS-Grade 1 or 2 Depth (wound above fascia without exposed muscle, tendon or bone); 2) DFU-wound area between 1-12cm2; 3) DFU-wound with or without clinical neuropathy; 4) DFU-wound lower extremity non-invasive Doppler studies with ankle-brachial index value ≥0.7 and/or Toe pressure ≥50mmHg; and, 5) without evidence of acute infection (e.g., cellulitis, abscess or osteomyelitis) at the time of enrollment.
* If the subject is a woman of childbearing potential she must be practicing an acceptable form of birth control, as determined by the Investigator. All females with an intact uterus must have a negative Beta-Human Chorionic Gonadotropin test (< 5mIU/mL) to proceed with study participation.

Exclusion Criteria:

* Any SC who is unable to provide written informed consent will not be enrolled for study participation.
* Any SC who is pregnant or breast feeding, will not be allowed to enroll, or continue, in the study, as pregnancy or breast feeding may impact the study results.
* Subjects with DFU-wounds less than 1cm-square or greater than 12cm-square will be excluded from the study.
* At the beginning of the four-week Screening Phase all SC will be scheduled for study-selected standard DFU wound treatment and off-loading of the study ulcer, as determined by the PI. Subject candidates who are unable to comply with the recommended off-loading of the selected DFU-study wound will be excluded from study.
* During the Screening Phase, any SC whose DFU wound demonstrates more than a fifty-percent (50%) reduction in wound area will be excluded from the study [37].
* Any SC with a current active history of alcohol or substance abuse will be excluded from study participation.
* Any SC receiving steroid therapy (prednisone), chemotherapy or biological therapies (e.g., Humira) within twelve-weeks will be excluded.
* Any SC with active cancerous lesions, with or without chemotherapy, will be excluded from study participation.
* Any SC having received hyperbaric oxygen therapy (HBOT) or the use of bioengineered skin substitutes (i.e., Dermagraft® or Apligraf®) within six-months will be excluded from study participation.
* Any SC receiving platelet-derived growth factor therapy (Regranex®, Ortho- McNeil) within six-months will be excluded from study participation.
* Any SC who is on dialysis (hemo- or peritoneal dialysis) or has end stage renal disease will be excluded from study participation.
* A SC with ABI values <0.7 or toe pressure <50mmHg, for the involved lower extremity of the study DFU-wound, will be excluded from study participation.
* A SC with a HgbA1C >9 will be excluded from study participation.
* Any SC with a medical condition, which, in the opinion of the investigator should exclude him/her from participating in the study.
* Any SC previously taking daily oral high-dose folic acid with B-vitamin supplements (HDFA; folic acid-5mg/cyanocobalamin- 4mg/pyridoxine-50mg) for DFU-wound treatment will not be considered for study participation until at least 28-days following the discontinuation of HDFA administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Measures of Wound Closure (actual and percentage) | 12 weeks
  Reduction of study wound areas
Number of Wounds with Complete Healing | 12 weeks
  Wounds with complete re-epithelialization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Boykin, MD, Principal Investigator — Hunter Holmes McGuire VAMC
Locations (1):
- Hunter Holmes McGuire VAMC, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No